CLINICAL TRIAL: NCT02716285
Title: Peppermint Oil for the Treatment of Irritable Bowel Syndrome: Optimizing Therapeutic Strategies Using Targeted Delivery
Acronym: PERSUADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL56000.068.16; METC162009; 2015-005467-16 (EudraCT Number)
Record Dates: First submitted 2016-03-08; First posted 2016-03-23 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Irritable Bowel Syndrome; Abdominal Pain; Colonic Diseases, Functional
Keywords: Irritable Bowel Syndrome; Abdominal pain; Targeted Delivery; Peppermint oil
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Colonic Diseases, Functional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ileocolonic release peppermint oil (Experimental): Colon-targeted-delivery capsule containing 182mg of Peppermint Oil, to be taken orally, 3 times daily for 8 weeks (first week, dosing will be titred).
  Interventions: Drug: Ileocolonic release peppermint oil
- Small intestinal release peppermint oil (Tempocol®) (Experimental): Enteric-coated capsule containing 182mg of Peppermint Oil that release the oil in the small intestine, to be taken orally, 3 times daily for 8 weeks (first week, dosing will be titred).
  Interventions: Drug: Small intestinal release peppermint oil
- Placebo (Placebo Comparator): Capsule containing microcrystalline cellulose, to be taken orally, 3 times daily for 8 weeks (first week, dosing will be titred).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ileocolonic release peppermint oil — Peppermint oil, menthae piperitae aetheroleum
  Arms: Ileocolonic release peppermint oil
Drug: Placebo — Placebo capsule, containing microcrystalline cellulose
  Arms: Placebo
Drug: Small intestinal release peppermint oil — Peppermint oil, menthae piperitae aetheroleum
  Other Names: Tempocol
  Arms: Small intestinal release peppermint oil (Tempocol®)

SUMMARY:
Peppermint oil has shown to be effective in the treatment of Irritable Bowel Syndrome (IBS) symptoms in several meta-analyses. However, the level of evidence is moderate and peppermint oil remains relatively under-used in IBS. Therefore, the investigators will conduct a multicenter randomized, placebo controlled trial to investigate the effects of an eight-week peppermint oil treatment in IBS patients according to current European Medicines Agency (EMA) / US Food and Drug Administration (FDA) guidelines. To improve efficacy and to reduce side effects, the investigators aim to study the use of a new peppermint oil formulation, a colon-targeted-delivery capsule that will release the oil in the (ileo-) colonic region specifically.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years;
2. Diagnosed with Irritable Bowel Syndrome according to the Rome IV criteria:

   (Recurrent abdominal pain, at least 1 day/week for the last 3 months; Symptom onset at least 6 months prior to diagnosis; Associated with two or more of the following:
   1. Pain related to defecation;
   2. Pain associated with a change in frequency of stool;
   3. Pain associated with a change in form (appearance/consistency) of stool
3. Based on the medical history and previous examination, no other causes for the abdominal complaints can be defined. Especially no history of:

   1. Inflammatory Bowel Disease;
   2. Celiac Disease;
   3. Thyroid dysfunction (if not well-regulated). If alarm symptoms (including unexplained rectal blood loss or weight loss) are present, a colonoscopy has been performed and was negative for other causes.
4. Women in fertile age (<55 years old) must use contraception or be postmenopausal for at least two years.
5. Average worst abdominal pain score (on 11-point NRS) of > 3, during the two-week run-in period.

Exclusion Criteria:

1. Insufficient fluency of the Dutch language;
2. Any previous use (also incidental use) of peppermint oil capsules in the last 3 months prior to inclusion (the use of peppermint tea, menthol candy etc. is allowed);
3. The inability to stop regular use of medication affecting the gastro-intestinal system (such as Non Steroidal Anti Inflammatory Drugs (NSAID), laxatives, prokinetics, opioids, smasmolytics and anti-diarrhoeal drugs). This use should be halted at least 1 week before enrollment into the run-in period;

   1. The use of 1 antidepressant drug is allowed, providing dosing has been stable for > 6 weeks before enrollment;
   2. The use of 1 proton pump inhibitor (PPI) is allowed, providing dosing has been stable > 6 weeks before enrollment;
4. Previous major abdominal surgery or radiotherapy interfering with gastrointestinal function:

   1. Uncomplicated appendectomy, cholecystectomy and hysterectomy allowed unless within the past 6 months;
   2. Other surgery upon judgment of the principle investigator;
5. History of liver disease, cholangitis, achlorhydria, gallstones or other diseases of the gallbladder/biliary system;
6. Pregnancy, lactation;
7. Using drugs of abuse;
8. Known allergic reaction to peppermint.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Abdominal pain response rate after 8 weeks of treatment | 8 weeks
  A responder is defined as a patient who experiences at least a 30 percent decrease in the weekly average of worst daily abdominal pain (measured daily, on an 11 point NRS) compared to baseline weekly average in at least 50 percent of the weeks in which the treatment in given.
Degree of relief response rate after 8 weeks of treatment. | 8 weeks
  A responder is defined as a patient who experiences a weekly relief of 1 or 2 (on a 7 point NRS) in at least 50 percent of the weeks in which treatment is given.

SECONDARY OUTCOMES:
Global symptom improvement | 8 weeks
  As determined by IBS-SSS (IBS symptom severity scale)
Abdominal Discomfort | 8 weeks
  As determined by symptom diary
Bloating | 8 weeks
  As determined by IBS-SSS (IBS - symptom severity scale)
Regurgitation | 8 weeks
  As determined by symptom diary
Nausea | 8 weeks
  As determined by symptom diary
Urgency | 8 weeks
  As determined by symptom diary
Abdominal cramps | 8 weeks
  As determined by symptom diary
Average stool frequency and consistency | 8 weeks
  Measured by bristol stool chart
Indirect costs | 8 weeks, 3 and 6 months
  Determined by Production Cost Questionnaire (PCQ) questionnaire
Direct costs | 8 weeks, 3 and 6 months
  Determined by Medical Cost Questionnaire (MCQ) questionnaire
General Quality of Life | 8 weeks, 3 and 6 months
  As determined by Euro-Qol-5D (EQ-5D)
IBS related Quality of Life | 8 weeks, 3 and 6 months
  As determined by IBS-Quality of life questionnaire (IBS-QoL)
Use of Over the counter medication and rescue medication | 8 weeks
  Number of drugs taken as rescue medication (This is not an intervention)
Number and severity of side effects | 8 weeks
  Determined by daily diary
Responder rates following discontinuation of treatment at 3 and 6 months, different thresholds for the responder analysis of abdominal pain (e.g. 40 and 50 percent improvement); | 3 and 6 months after discontinuation of treatment
Responder rates when missing are interpreted as "no effect" | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A Masclee, Prof., PhD., MD., Principal Investigator — Maastricht University Medical Center
Locations (4):
- Netherlands (4):
  - Gelderse Vallei Hospital, Ede, Gelderland
  - Medical Center Leeuwarden, Leeuwarden, Provincie Friesland
  - Alrijne Hospital, Leiden, South Holland
  - Maastricht University Medical Center, Maastricht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schellekens RC, Stellaard F, Olsder GG, Woerdenbag HJ, Frijlink HW, Kosterink JG. Oral ileocolonic drug delivery by the colopulse-system: a bioavailability study in healthy volunteers. J Control Release. 2010 Sep 15;146(3):334-40. doi: 10.1016/j.jconrel.2010.05.028. Epub 2010 May 31. PMID 20621586
- [Background] Maurer JM, Schellekens RC, van Rieke HM, Stellaard F, Wutzke KD, Buurman DJ, Dijkstra G, Woerdenbag HJ, Frijlink HW, Kosterink JG. ColoPulse tablets perform comparably in healthy volunteers and Crohn's patients and show no influence of food and time of food intake on bioavailability. J Control Release. 2013 Dec 28;172(3):618-24. doi: 10.1016/j.jconrel.2013.09.021. Epub 2013 Oct 2. PMID 24096020
- [Background] Khanna R, MacDonald JK, Levesque BG. Peppermint oil for the treatment of irritable bowel syndrome: a systematic review and meta-analysis. J Clin Gastroenterol. 2014 Jul;48(6):505-12. doi: 10.1097/MCG.0b013e3182a88357. PMID 24100754
- [Background] Enck P, Junne F, Klosterhalfen S, Zipfel S, Martens U. Therapy options in irritable bowel syndrome. Eur J Gastroenterol Hepatol. 2010 Dec;22(12):1402-11. doi: 10.1097/MEG.0b013e3283405a17. PMID 21389791
- [Background] Ford AC, Talley NJ, Spiegel BM, Foxx-Orenstein AE, Schiller L, Quigley EM, Moayyedi P. Effect of fibre, antispasmodics, and peppermint oil in the treatment of irritable bowel syndrome: systematic review and meta-analysis. BMJ. 2008 Nov 13;337:a2313. doi: 10.1136/bmj.a2313. PMID 19008265
- [Background] Weerts ZZRM, Keszthelyi D, Vork L, Aendekerk NCP, Frijlink HW, Brouwers JRBJ, Neef C, Jonkers DMAE, Masclee AAM. A Novel Ileocolonic Release Peppermint Oil Capsule for Treatment of Irritable Bowel Syndrome: A Phase I Study in Healthy Volunteers. Adv Ther. 2018 Nov;35(11):1965-1978. doi: 10.1007/s12325-018-0802-1. Epub 2018 Oct 4. PMID 30284674
- [Derived] Weerts ZZRM, Essers BAB, Jonkers DMAE, Willems JIA, Janssen DJPA, Witteman BJM, Clemens CHM, Westendorp A, Masclee AAM, Keszthelyi D. A trial-based economic evaluation of peppermint oil for the treatment of irritable bowel syndrome. United European Gastroenterol J. 2021 Nov;9(9):997-1006. doi: 10.1002/ueg2.12134. Epub 2021 Sep 1. PMID 34468079
- [Derived] Weerts ZZRM, Masclee AAM, Witteman BJM, Clemens CHM, Winkens B, Brouwers JRBJ, Frijlink HW, Muris JWM, De Wit NJ, Essers BAB, Tack J, Snijkers JTW, Bours AMH, de Ruiter-van der Ploeg AS, Jonkers DMAE, Keszthelyi D. Efficacy and Safety of Peppermint Oil in a Randomized, Double-Blind Trial of Patients With Irritable Bowel Syndrome. Gastroenterology. 2020 Jan;158(1):123-136. doi: 10.1053/j.gastro.2019.08.026. Epub 2019 Aug 27. PMID 31470006